CLINICAL TRIAL: NCT05520073
Title: A Feasibility Study for Decentralized Clinical Trial: an Open-label, Randomized, Remote Clinical Trial to Evaluate the Effects of Lactobacillus Supplements on Alleviating Functional Constipation Symptoms in Poor-health Volunteers
Brief Title: A Pilot Study To Evaluate the Effects of Lactobacillus Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kyung-Sang Yu, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DCT-101
Record Dates: First submitted 2022-08-24; First posted 2022-08-29 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Feasibility Studies
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactobacillus and Vitamin C (Experimental): Lactobacillus and Vitamin C supplements daily self-administration for 14 days
  Interventions: Dietary Supplement: Lactobacillus plantarum; Dietary Supplement: Vitamin C
- Vitamin C (Placebo Comparator): Vitamin C supplements daily self-administration for 14 days
  Interventions: Dietary Supplement: Vitamin C

INTERVENTIONS:
Dietary Supplement: Lactobacillus plantarum — Lactobacillus product 1 pack daily
  Arms: Lactobacillus and Vitamin C
Dietary Supplement: Vitamin C — Vitamin C tablet 1 pack daily

SUMMARY:
This is a feasibility study to evaluate a decentralized (remote) clinical trial in Korea. In this study, an open-label, randomized, remote clinical trial to evaluate the effects of lactobacillus supplements on alleviating functional constipation symptoms in poor-health volunteers will be conducted.

DETAILED DESCRIPTION:
This study was designed for the purpose of confirming the feasibility of conducting a distributed clinical trial in the domestic medical environment and practically checking the considerations during implementation. This clinical trial aims to evaluate the effectiveness of interventions for functional constipation, a chronic disease, through the design of a fully distributed clinical trial, which is the most advanced form of distributed clinical trial. There are many patients with functional constipation around the world, and the need for a comparative randomized clinical trial for new treatments is being emphasized. It is expected to have a high potential for use in that it can be evaluated as In particular, health functional food preparations such as lactobacillus preparations have been reported to have effects on functional constipation, but it is difficult to prove their effectiveness due to the heterogeneity of clinical trial design5, so it can be considered as an application field for distributed clinical trials.

For this purpose, we intend to try an exploratory clinical trial to evaluate the effectiveness of lactic acid bacteria preparations in a distributed environment. In this clinical trial, patients are recruited remotely through a website, and visits to medical institutions are minimized by delivering lactic acid bacteria to home delivery and evaluating symptom improvement through self-recording symptoms. In addition, it is intended to ensure the accuracy of the collected data by having the urine vitamin C test be performed by oneself to check whether the drug is administered or not. Through this, it is expected that issues and considerations that may arise when designing distributed clinical trials in the future can be derived.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 19 and 64 years
* In the past 6 months, one or more of the following symptoms have been present for at least 2 weeks without having to be consecutive (based on alleviated Rome III functional constipation)

  1. Excessive strain during defecation exceeds 1/4 of the total number of bowel movements
  2. Lumpy or hard stool exceeds 1/4 of the total number of bowel movements
  3. Feeling after defecation exceeds 1/4 of the total number of bowel movements
  4. The feeling of anal obstruction during defecation exceeds 1/4 of the total number of bowel movements
  5. More than 1/4 of the total number of bowel movements that require manual manipulation to help defecate
  6. Less than 3 bowel movements per week
* A person who voluntarily decides to participate after hearing and fully understanding the detailed explanation of this clinical trial and consents before screening

Exclusion Criteria:

* Those who have a clinically significant hypersensitivity reaction to lactic acid bacteria, vitamin C, or ingredients included in the drug
* Persons with a history or evidence of clinically significant blood, renal, endocrine, respiratory, gastrointestinal, urinary, cardiovascular, liver, psychiatric, neurological or immune disease (eg, colorectal cancer, etc.)
* Those who are pregnant or lactating
* Those who cannot faithfully record self-recording of dosing and defecation within the clinical trial period
* Those who are taking or expected to take lactic acid bacteria or vitamin C preparations other than health functional foods to be administered in clinical trials within the period from 2 weeks before the scheduled first dose to the last dose
* Those who judged that the investigator is inappropriate to participate in the clinical trial due to other reasons

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Frequency of spontaneous defecation | 21 days
  Frequency of spontaneous defecation
Formation of stool | 21 days
  According to Bristol Stool Scale
Other symptoms related to defecation | 21 days
  e.g. Excessive straining, bloating, anal obstruction, abdominal pain and discomfort, and manipulation of the fingers

OTHER OUTCOMES:
The number of days on which self-records were made among the scheduled 21 days | 21 days
  Feasibility assessment for DCT elements
Completeness of self-record | 21 days
  Feasibility assessment for DCT elements
Number of times self-records were written on the due date | 21 days
  Feasibility assessment for DCT elements
The proportion of completed of dosing and defecation record | 21 days
  Feasibility assessment for DCT elements
Proportion of the positive and negative opinions on the overall DCT procedures | 21 days
  Feasibility assessment for DCT elements

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital Clinical Trial Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No